CLINICAL TRIAL: NCT05234944
Title: A Brief Telehealth Intervention to Address Diabetes Health-related Quality of Life (HRQOL) in Families of Youth and Adults with Type 1 Diabetes Across Clinical Settings: a Pilot and Feasibility Study
Brief Title: Pilot Study of Brief Intervention to Support Diabetes Health-Related Quality of Life
Acronym: T1DALPilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Marisa Hilliard, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-50359
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: behavioral intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Non-randomized pilot study, all participants will receive intervention
Masking Description: Non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): A CDCES trained by the research team will deliver the intervention via HIPAA compliant telehealth/videoconferencing platform. There will be 2 sessions within approximately 6 months. Prior to each session, participants will complete an assessment of T1D-specific health-related quality of life, which will generate a summary report for each person that lists aspects of quality of life that are going well and aspects that are potential areas for improvement. The CDCES will review the reports with the participants, focusing on building on areas of strength and teaching brief behavioral strategies or resources to address aspects of quality of life that could be improved. Strategies may include stress management, problem-solving techniques, goal-setting, strategies to seek social support, or other brief behavioral skills. The CDCES will also offer information about relevant resources and will provide referrals for mental health support as needed.
  Interventions: Behavioral: Type 1 Diabetes and Life

INTERVENTIONS:
Behavioral: Type 1 Diabetes and Life — Brief behavioral intervention, delivered remotely by certified diabetes care and education specialists, targeting diabetes-specific health-related quality of life for people with type 1 diabetes across the lifespan and for their parents and partners.

SUMMARY:
The aims of this pilot study are to evaluate the feasibility, acceptability, preliminary impact, and costs of a brief, behavioral intervention delivered remotely by diabetes educators to people with type 1 diabetes and their family members. The purpose of the intervention is to support health-related quality of life for people with type 1 diabetes of all ages and to support the diabetes health-related quality of life of their parents and partners. This pilot study will explore how this intervention works as a supplement to routine medical care in three clinical care settings: an adult specialty diabetes care setting, a pediatric subspecialty diabetes care setting, and for people who receive diabetes medical care from a primary care provider. To maximize data about feasibility and acceptability of the intervention, all participants in the pilot study will receive the intervention and there will not be randomization to a control condition.

DETAILED DESCRIPTION:
The aims of this pilot study are to evaluate the feasibility, acceptability, preliminary impact, and costs of a brief behavioral intervention to support diabetes health-related quality of life, delivered remotely by diabetes educators to people with type 1 diabetes and their family members. The key components of the intervention include people with diabetes and their parents/partners completing a validated measure of diabetes-specific health-related quality of life around the time of two consecutive diabetes clinic appointments. A trained study certified diabetes care and education specialist (CDCES) will meet remotely (via secure, HIPAA-compliant cloud-based telehealth/videoconferencing platform) to guide the family in a brief discussion about each person's diabetes health-related quality of life. They will discuss the parts of quality of life that are going well and the parts that are more challenging, and the CDCES will teach brief behavioral strategies to address quality of life challenges. Using a non-randomized design, all participants will receive the intervention for the pilot study. Participants will complete surveys prior to receiving the intervention and again after the completion of the intervention, and clinical data will be collected from the person with diabetes and their medical records.

To evaluate this pilot intervention, the specific aims are: (1) Evaluate the feasibility and acceptability of the intervention for participants in three clinical settings: pediatric subspecialty clinic, adult specialty clinic, and diabetes care from primary care providers. (2) Examine preliminary indicators of pre-post change in behavioral and clinical outcomes. (3) Explore costs associated with intervention delivery and receipt to inform the next phases of intervention development and testing.

ELIGIBILITY:
Inclusion Criteria (People with Diabetes):

* Type 1 diabetes diagnosis for at least 12 months
* Treated at the participating clinical site (for the pediatric and adult subspecialty sites)
* Fluent in English

Inclusion Criteria (Parents/Partners):

* Age 18 years or older.
* Child/Partner with diabetes participating in study
* Fluent in English

Exclusion Criteria (all participants):

* Any major comorbid medical (PWD only), cognitive, or psychiatric condition that would limit ability to participate
* Plans to move to another clinical site during the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of participant accrual, data collection, intervention delivery | Post-intervention, up to 6 months
  Feasibility of conducting a research study about this intervention will be measured by percentage of eligible participants who consent to the study, complete questionnaires, and receive the full intervention dose. These outcomes will be calculated based on recruitment and program delivery tracking conducted by study staff
Acceptability | Post-intervention, up to 6 months
  Participants will complete brief surveys at study completion that assess their experiences with the intervention, including helpfulness of conversations, value of time spent, overall acceptability of program, and recommendations for improvement. Items will be rated using a Likert-scale, with higher scores indicating higher satisfaction with each item.

SECONDARY OUTCOMES:
Diabetes health-related quality of life | Baseline and Post-intervention, up to 6 months
  Participants will complete the age- and respondent-appropriate version of the Type 1 Diabetes and Life (T1DAL) measure. Psychometric data regarding the validity and reliability of the pediatric, adult, and parent/partner versions of the T1DAL are published. Total scores are on a 100-point scale, with higher scores indicating better quality of life.
  This is the only measure that will also be collected at the mid-point (before 2nd visit) between the two intervention sessions. Participant responses on the baseline and midpoint T1DAL measures will be automatically scored (per an algorithm designed by the study investigator team) and used to generate a quality of life profile that the CDCES will use in each intervention session.
Diabetes distress | Baseline and Post-intervention, up 6 months
  Participants will complete the age- and respondent-appropriate version of the Problem Areas in Diabetes (PAID) scale (children, adolescents, and parents) or the Diabetes Distress Scale (adults and partners). Higher scores on each measure indicate more distress.
Adherence/Diabetes Self-management | Baseline and Post-intervention, up to 6 months
  Participants will complete the Self-Care Inventory Revised. Higher scores indicate higher adherence/more engagement in diabetes self-management behaviors. For youth under age 12, parents will complete this measure about the child's self-management behaviors because this measure has not been validated for self-report use by children. Parents of youth age 12 or older and partners of adults will not complete any measures of self-management behavior.
Glycemic Outcome - HbA1c | Baseline and Post-intervention, up to 6 months
  Point of care HbA1c values documented by the medical team at each clinic visit during which an intervention session takes place, plus the following clinic visit (3-6 months after the second intervention session) will be collected from the electronic health record, to assess change in glycemic outcomes. For participants in the primary care group, participants will self-report the date and value of their most recent HbA1c at each time point. They will be asked to upload a photo/PDF of documentation of their HbA1c value (e.g., lab results printout) if available. Participants in the primary care group will also be asked to complete a research home fingerstick HbA1c kit. Higher HbA1c indicates higher average blood glucose values over the previous 2-3 months, which represents poorer glycemic control.
Glycemic Outcome - Time in Range | Baseline and Post-intervention, up to 6 months
  When available for participants who use a continuous glucose monitor (CGM), 14 days' of CGM data will be downloaded at each time point by the study teams to calculate glucose time-in-range as an additional index of glycemic control. Higher time-in-range is an indicator of better glycemic control.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Hilliard, PhD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Joslin Diabetes Center at SUNY Upstate Medical University, Syracuse, New York
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share de-identified data for all IPD that underlie results in a publication on request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication
Access Criteria: Upon request to PI